CLINICAL TRIAL: NCT05436210
Title: The Impact of Postural and Anthropometric Properties of Foot and Ankle on Physical Performance and Ambulation of Patients With Duchenne Muscular Dystrophy
Brief Title: Postural and Anthropometric Properties of Foot and Ankle of Patients With DMD
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Güllü AYDIN YAĞCIOĞLU, Principal Investigator, Hacettepe University
Other Study IDs: GO 22/414
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Duchenne Muscular Dystrophy; Ambulation Difficulty; Posture Disorders in Children; Ambulation Disorder, Neurologic
Keywords: Duchenne Muscular Dystrophy; foot posture; performance; ambulation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Mobility Limitation; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: foot posture index, north star ambulation assessment, timed performance tests, 6 minute walk test — Patients will be evaluated only observationally without intervention by foot posture index, north star ambulation assessment, timed performance tests, 6 minute walk test

SUMMARY:
Introduction: Progressive muscle weakness, joint contractures and body alignment disorders seen in patients with Duchenne Muscular Dystrophy (DMD) adversely affect the foot structure of the patients.

Objective: The aim of this study is to examine the relationship between foot posture, performance and ambulation in patients with DMD.

Method: The patient with ambulatory DMD will be included in the study. The foot postures of the patients will be evaluated with the Foot Posture Index. Relationships between the Foot Posture Index and performance tests (6 minute walk test, timed performance tests (10m walking, Gower's, climb/descend 4 stair)) and the North Star Ambulation Evaluation, an ambulation evaluation, will be examined.

ELIGIBILITY:
Inclusion Criteria:

1.5 to 18 years old 2. Not to have lost his ambulation 3. Agreeing to participate in the research voluntarily

Exclusion Criteria:

1. Having serious mental and psychological problems,
2. Having lost his ambulation
3. Inability to cooperate adequately with the physiotherapist who made the evaluations,
4. Any injury and/or surgery to the lower extremities in the last 6 months.

Ages: 5 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ambulated Duchenne Muscular Dystrophy patients aged of 5-18 years
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
foot posture index - 6 | 10 minutes
  The Foot Posture Index - 6 (FPI-6) was evaluated with each child standing and using the original protocol. FPI-6 values ranged from -2 to +2 for each of the six criteria and from -12 to +12 for the total score, indicative of position of each foot along the supinated to pronated continuum of foot posture.
6 min walk test (6MWT) | 6 minutes
  Six Minute Walk Test was used commonly in DMD were found to be valid, reliable and easy to apply in the clinic. Children were asked to walk during 6 minutes as fast as they can at a corridor specified by two cones and walking distances were recorded as meter (m) for 6MWT. The time passed during timed performance tests were recorded as seconds.
north star ambulation assessment | 10 minutes
  Patients' ambulation will be evaluated with the North Star Ambulation Assessment (NSAA). The NSAA consists of 17 items and evaluates ambulation with functional activities such as walking, getting up from a chair, going up and down stairs, and running. Each item is scored in the range of 0-2 points and the total score is in the range of 0-34. High score indicates better ambulation status
timed performance test | ten minutes
  Ascending-descending standard 4 steps, walking 10m, standing from lying position were used in order to assess the performance of children.The time passed during timed performance tests were recorded as seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Güllü Aydın Yağcıoğlu, Isparta, Turkey (Türkiye)